CLINICAL TRIAL: NCT06455111
Title: Evaluation of an Artificial Intelligence-Assisted, Image-Based Dietary Assessment Tool in the Framingham Heart Study: A Block Randomized Controlled Trial
Brief Title: Evaluation of an Artificial Intelligence-Assisted, Image-Based Dietary Assessment Tool in the Framingham Heart Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-41743; R01DK129305 (NIH)
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Dietary Habits
Keywords: Web-based dietary recalls; Automatic Self-Administered 24-Hour Dietary Assessment Tool; Keenoa; Framingham Heart Study cohort
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: A randomized block design will be implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keenoa (Experimental): Participants randomized to this arm will document a 3-day dietary assessment using Keenoa.
  Interventions: Other: Keenoa
- ASA24 (Active Comparator): Participants randomized to this arm will document a 3-day dietary assessment using the web-based Automatic Self-Administered 24-Hour (ASA24) Dietary Assessment Tool.
  Interventions: Other: ASA24

INTERVENTIONS:
Other: Keenoa — Keenoa is an artificial intelligence-enhanced, image-assisted tool, is a newly designed mobile application that may facilitate collection of dietary data. Serving as a visual food diary, individuals can upload a picture of their meal, choose the food items eaten using a preselected food list available by the app, and confirm the portion size with the presented visual aids.
  Arms: Keenoa
Other: ASA24 — The Automated Self-Administered 24-Hour (ASA24) dietary recall or record is a free, web-based tool that enables multiple, automatically coded, self-administered 24-hour diet recalls and/or single or multi-day food records, also known as food diaries.
  Arms: ASA24

SUMMARY:
Assessment of dietary intake in large, free-living populations is inherently challenging due to the complex nature of human diet. Advancements in traditional methods of dietary assessment (i.e., web-based dietary recalls or records) have aimed at improving data accuracy while reducing participant burden. Further utilizing food recognition technologies to capture real-time food intake may aid in overcoming limitations of existing methods. Keenoa, an artificial intelligence-enhanced, image-assisted tool, is a newly designed mobile application that may facilitate collection of dietary data.

Primarily, the investigators will assess acceptability and usability of Keenoa compared with the traditional, web-based Automatic Self-Administered 24-Hour (ASA24) Dietary Assessment Tool in the Framingham Heart Study Third Generation-based cohorts at examination 4. The investigators will also determine the proportion of participants who complete all three days of dietary assessment, either through Keenoa or ASA24. Further, the investigators will relate dietary determinants of glycemic variability (e.g., percent carbohydrate, fiber intake, etc.), obtained from each dietary assessment tool, to the continuous glucose monitor (CGM)-derived outcomes.

With a randomized block design, this study will take place as part of the Framingham Heart Study (FHS) glucose study (R01 DK129305). Currently participants from the Third Generation-based cohorts are asked at their fourth examination to wear Dexcom G6 Pro continuous glucose monitor on either their arm or abdomen for a duration of at least 4 days. During this time, participants are asked to complete 3 consecutive days of dietary record through ASA24. For this trial, the investigators will randomize the dietary assessment tool weekly between ASA24 and Keenoa, therefore, depending on the week of administration, participants will be randomized to either a 3 days dietary record via ASA24 or a 3-day dietary record through Keenoa. This trial will last a total of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* FHS participants from the Gen 3 cohort who will attend the Exam 4 cycle

Exclusion Criteria:

* Participants with cognitive impairment which may prevent them from being able to complete diet records and follow instructions for continuous glucose monitor device wear.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole L Spartano, PhD, Principal Investigator — BU Chobanian & Avedisian School of Medicine
Locations (1):
- BU Chobanian & Avedisian School of Medicine, Framingham Heart Study, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Keenoa | ASA24
Started | 64 | 51
Completed | 53 | 47
Not Completed | 11 | 4
Not completed — Withdrawal by Subject | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Keenoa | ASA24 | Total
Number analyzed (Participants) | 64 | 51 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (7.9) | 58.4 (9.0) | 58.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 27 | 62
  Male | 29 | 24 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hon-Hispanic White | 59 | 47 | 106
  Non-Hispanic Black | 1 | 0 | 1
  Non-Hispanic Multiracial | 2 | 1 | 3
  Non-Hispanic Unknown Race | 0 | 1 | 1
  Hispanic/Latino | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 64 | 51 | 115

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Dietary Assessment Method
Description: Acceptability will be assessed using a quantitative satisfaction scale (0-5), where 0=not acceptable and 5=very acceptable. Higher scores suggest higher acceptability.
Time Frame: 6 weeks
Population: 38 participants in the Keenoa group and 27 participants in the ASA24 group provided answers about acceptability used to analyze this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Keenoa | ASA24
Number analyzed (Participants) | 38 | 27
units on a scale | 3.3 (1.1) | 3.1 (0.99)

2. Primary Outcome: Completion of 3 Day Dietary Assessment With >= 600 kcal
Description: This outcome will be assessed by the number and percentage of participants who complete all 3 days of diet assessments with >= 600 kcal. The higher the percentage the greater the completion rate.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Keenoa | ASA24
Number analyzed (Participants) | 53 | 47
Participants | 23 | 27

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Keenoa | ASA24
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/47
Other Adverse Events (participants affected / at risk) | 0/53 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT06455111/Prot_SAP_001.pdf
  • Informed Consent Form (2024-04-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT06455111/ICF_000.pdf